CLINICAL TRIAL: NCT00278213
Title: Consolidation With Campath-1H After FMC Induction in Patients With T-cell Chronic Lymphocytic Leukemia
Brief Title: Combination Chemotherapy Followed By Alemtuzumab in Treating Patients With Chronic Lymphocytic Leukemia or Prolymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: German CLL Study Group (Other)
Masking: None | Purpose: Treatment
Other Study IDs: T-PLL1; EU-20562
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Prolymphocytic Leukemia
Keywords: prolymphocytic leukemia; refractory chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; T-cell large granular lymphocyte leukemia
MeSH Terms: conditions — Leukemia, Prolymphocytic; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Large Granular Lymphocytic | interventions — Alemtuzumab; Cyclophosphamide; fludarabine phosphate; Mitoxantrone

INTERVENTIONS:
Biological: alemtuzumab
Drug: cyclophosphamide
Drug: fludarabine phosphate
Drug: mitoxantrone hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fludarabine, cyclophosphamide, and mitoxantrone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells. Monoclonal antibodies, such as alemtuzumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others can find cancer cells and help kill them or carry cancer-killing substances to them. Combination chemotherapy followed by alemtuzumab may be effective in treating chronic lymphocytic leukemia and prolymphocytic leukemia.

PURPOSE: This phase II trial is studying how well giving combination chemotherapy followed by alemtuzumab works in treating patients with T-cell chronic lymphocytic leukemia or prolymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the number of severe adverse events and life-threatening infections in patients with T-cell chronic lymphocytic leukemia or T-cell prolymphocytic leukemia treated with induction chemotherapy comprising fludarabine, cyclophosphamide, and mitoxantrone hydrochloride followed by consolidation therapy comprising alemtuzumab.
* Determine the remission rate in patients treated with this regimen.

Secondary

* Determine the overall and progression-free survival of patients treated with this regimen.
* Determine the quality of remission in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive induction chemotherapy comprising fludarabine IV and cyclophosphamide IV for 3 days and mitoxantrone hydrochloride IV on 1 day. Treatment repeats every 28 days for up to 4 courses. Patients then receive consolidation therapy comprising alemtuzumab IV 3 times in week 1 and then weekly for up to 11 weeks.

PROJECTED ACCRUAL: A total of 17 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of T-cell chronic lymphocytic leukemia (T-CLL) or T-cell prolymphocytic leukemia (T-PLL)
* Previously untreated disease OR patient may have received up to 2 therapies

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 6 months
* No severe organ dysfunction
* No other concurrent or previous neoplasm
* No autoimmune hemolytic anemia or thrombocytopenia

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior fludarabine, mitoxantrone hydrochloride, cyclophosphamide, or alemtuzumab

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2002-09; Primary Completion 2007-02 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Adverse effects at 2 months after treatment
Remission rate at 2 months after treatment

SECONDARY OUTCOMES:
Overall survival at 2 months after treatment
Progression-free survival at 2 months after treatment
Remission quality at 2 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Georg Hopfinger, Study Chair — Hanusch-Krankenhaus
Locations (19):
- Austria (2):
  - Allgemeines Krankenhaus - Universitatskliniken, Vienna
  - Hanuschkrankenhaus, Vienna
- Germany (17):
  - Allgemeinen Krankenhaus Celle Kinderklinik, Celle
  - St. Johannes Hospital - Medical Klinik II, Duisburg
  - Helios Klinikum Erfurt, Erfurt
  - Universitaetsklinikum Essen, Essen
  - Klinikum Garmisch - Partenkirchen GmbH, Garmisch-Partenkirchen
  - Sana Klinikum Hof, Hof
  - University Hospital Schleswig-Holstein - Kiel Campus, Kiel
  - Internistische Praxis - Ludwigsburg, Ludwigsburg
  - Sana Kliniken Luebeck, Lübeck
  - Haematologische Praxis - Moenchengladbach, Mönchengladbach
  - Gemeinschaftliche Schwerpunktpraxis - Osnabrueck, Osnabrück
  - Schwerpunktpraxis fuer Haematologie und Onkologie, Saarbrücken
  - Caritasklinik St. Theresia, Saarbrücken
  - Southwest German Cancer Center at Eberhard-Karls-University, Tübingen
  - Dr. Horst-Schmidt-Kliniken, Wiesbaden
  - Hamatologisch - Onkologische Praxis Wurzburg, Würzburg
  - Klinikum des Landkreises Loebau-Zittau GmbH, Zittau

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hopfinger G, Busch R, Pflug N, Weit N, Westermann A, Fink AM, Cramer P, Reinart N, Winkler D, Fingerle-Rowson G, Stilgenbauer S, Dohner H, Kandler G, Eichhorst B, Hallek M, Herling M. Sequential chemoimmunotherapy of fludarabine, mitoxantrone, and cyclophosphamide induction followed by alemtuzumab consolidation is effective in T-cell prolymphocytic leukemia. Cancer. 2013 Jun 15;119(12):2258-67. doi: 10.1002/cncr.27972. Epub 2013 Mar 19. PMID 23512246